CLINICAL TRIAL: NCT00005351
Title: Incidence and Outcomes of Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4226; R01HL046974 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2002-09

CONDITIONS: Cardiovascular Diseases; Lung Diseases; Pulmonary Embolism; Venous Thromboembolism
MeSH Terms: conditions — Cardiovascular Diseases; Lung Diseases; Pulmonary Embolism; Venous Thromboembolism

SUMMARY:
To identify the incidence cohort of Olmsted County Minnesota residents with deep venous thrombosis (DVT)/pulmonary embolism (PE) from 1966 through 1990. Episodes of DVT or PE acquired during hospitalization or in the community were identified for future studies.

DETAILED DESCRIPTION:
BACKGROUND:

Deep vein thrombosis and pulmonary embolism most often occur during hospitalization for surgery or chronic medical conditions. Consequently information on deep venous thrombosis/pulmonary embolism is derived from large referral hospitals, and there are substantial gaps in our understanding of the incidence, risk factors, and outcomes of deep venous thrombosis/pulmonary embolism in the community. This was one of the first studies to compare hospital acquired deep venous thrombosis/pulmonary embolism with deep venous thrombosis/pulmonary embolism among ambulatory residents in a community.

DESIGN NARRATIVE:

The five part study: 1. identified the incidence cohort and tested the hypotheses that over the 25 year study period the incidence of deep venous thrombosis/pulmonary embolism had decreased, the extent of testing for suspected deep venous thrombosis/pulmonary embolism had increased, and the number of tests obtained for patients with deep venous thrombosis/pulmonary embolism had increased. 2. determined the independent risk factors for deep venous thrombosis/pulmonary embolism and estimated the population attribute risk due to each independent risk factor for deep venous thrombosis/pulmonary embolism in a case-control study of the incidence cohort and community controls. 3. tested the hypothesis that deep venous thrombosis/pulmonary embolism were independent risk factors for death after adjusting for age, sex and co-morbid conditions. 4. described the occurrence of the post-phlebitic syndrome, pulmonary hypertension, and recurrent deep venous thrombosis/pulmonary embolism over the 25 year study period and identified the independent risk factors for lower extremity venous ulceration. 5. evaluated the accuracy of national pulmonary embolism mortality rates by comparing pulmonary embolism mortality rates calculated from a review of all the inpatient and outpatient medical records of Olmsted County deep venous thrombosis/pulmonary embolism patients with death certificate pulmonary embolism mortality rates for Olmsted County from the National Center for Health Statistics. The study provided the most complete and comprehensive population based estimates of the incidence, risk factors, survival and outcomes of deep venous thrombosis/pulmonary embolism available to date.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-08; Study Completion 1994-07 (Actual)

REFERENCES:
- [Background] Silverstein MD, Heit JA, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ 3rd. Trends in the incidence of deep vein thrombosis and pulmonary embolism: a 25-year population-based study. Arch Intern Med. 1998 Mar 23;158(6):585-93. doi: 10.1001/archinte.158.6.585. PMID 9521222
- [Background] Gitter MJ, Jaeger TM, Petterson TM, Gersh BJ, Silverstein MD. Bleeding and thromboembolism during anticoagulant therapy: a population-based study in Rochester, Minnesota. Mayo Clin Proc. 1995 Aug;70(8):725-33. doi: 10.4065/70.8.725. PMID 7630209